CLINICAL TRIAL: NCT01335243
Title: Multicentric, Prospective Study of Efficacy and Safety of Lumbar Interbody Fusion With MatriTMBONE Associated With Autologous Marrow
Brief Title: Efficacy and Safety Study of Lumbar Interbody Fusion With MatriTMBONE Associated With Autologous Bone Marrow
Acronym: MatriBone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/21
Record Dates: First submitted 2011-04-06; First posted 2011-04-14 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Degenerative Osteoarthritis; Degenerative Lumbar Vertebra
Keywords: Orthopedic Procedures; Spine; Interbody fusion; Arthrodesis; Lumbar Vertebrae; CT Scan; Spine balance; Instrumented fusion; Posterior fusion; Degenerative spine; painful
MeSH Terms: conditions — Joint Diseases; Ankylosis; Pain | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TLIF surgery (Experimental)
  Interventions: Procedure: The Transforaminal Lumbar Interbody Fusion (TLIF) surgery

INTERVENTIONS:
Procedure: The Transforaminal Lumbar Interbody Fusion (TLIF) surgery — The TLIF surgery use a per-operating artificial substitute specific biomaterial: autologous osteoblasts punctured on iliac crest and put on a collagen support waxed with tri-calcium phosphate (which is osteoconductive) to perform a intervertebral body fusion.

SUMMARY:
The main objective of this clinical study is the estimation of the rate of intersomatic fusion observed 12 months after lumbar interbody fusion by posterior approach with PEEK interbody cage of fusion in PEEK performed with autologous bone of decortication and osseous substitute with a biomaterial (MatriBONE associated with the autologous bone marrow), associated with a posterolateral bone graft performed with MatriBone waxed with bone marrow. Indication is dedicated for patients by painful degenerative osteoarthritis, by narrow lumbar canal and\or spondylolisthesis.

DETAILED DESCRIPTION:
This clinical study corresponds to a TLIF surgery using a per-operating artificial substitute specific biomaterial: autologous osteoblasts punctured on iliac crest and put on a collagen support waxed with tri-calcium phosphate (which is osteoconductive) to perform a intervertebral body fusion.

Biomaterial MATRITM BONE: Device of class III, with marking IT in the indication of arthrodesis. It will be administered during the lumbar interbody fusion's procedure.

The material is a matrix of collagen mineralized containing a homogeneous mixture of collagen cleansed of type I+III and an osseous biphasic substitute HA / TCP. The proportion of both constituents is 90 % of osseous substitute for 10 % of collagen en masse. The collagen is reduced in approximately 1 month and the osseous substitute leads to an osseous reshaping in 6 - 9 months approximately.

The follow up will last 12 months with 2 visits (6 and 12 months after surgery), 2 CT scan slides before inclusion and at 12 months, classical X-rays before inclusion and at 6 and 12 months, questionnaires (visual analogic scale for pain, and quality of life with OSWESTRY and SF36 scales) before inclusion and at 6 and 12 months, and biological exams (CRP/VS, for inflammation) at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years old.
* Body mass index lower than 35
* Degenerative osteoarthritis painful and invalidating degenerative lumbar vertebra for at least 6 months and resistance fighter in the conservative treatment
* Narrow lumbar canal and\or spondylolisthesis with neurological disorder associated with signs of primary instability or induced to neurological liberation
* Patient requiring a surgery on a single interbody level.
* Given informed consent
* Patient with French health system

Exclusion Criteria:

* For women: no efficient contraception (intra uterine device, or contraceptive pill)
* Pregnant or feeding women
* Surgery zone local infection local
* Lumbar interbody fusion of more than two levels
* Spondylolisthesis of high rank (stage 3 or 4 of the classification of Meyerding)
* Scoliosis lumbar vertebra gives a complex to (Cobb angle> 40°)
* All surgical contraindications
* Severe hyperparathyroidism: calcium > 2,45 mmol/l and [PTH] ≥ 50pg / ml
* Uncontrolled diabetes (untreated or non stabilized by treatment)
* Long corticoid treatment (more than 6 months and stopped since less than 3 months)
* Current Chemotherapy or during the last three months
* Antecedent of regional radiotherapy
* All contraindication to MatriTM BONE: osteomyelitis, bone degenerative disease or necrosis of surgery site.
* Known turned out Osteoporosis untreated (dexa: > 2 DS)
* Subject participating in another research including a period of always current exclusion in the pre-inclusion
* Person placed under protection of justice
* Severely altered physical and\or psychological Health, which according to, the investigator, can affect to participant's compliance to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
patients' proportion which an intervertebral fusion | 12 months
  The main assessment criteria of this study are patients' proportion which an intervertebral fusion is documented to CT scanners The intervertebral fusion is documented by the revealing of at least an osseous continuous span of a vertebral level in the other one on one of three CT scan slides centred on the cage.

SECONDARY OUTCOMES:
NOTION OF TOLERANCE: Frequency and gravity of unwanted Adverse Events linked to the procedure and\or the use of the biomaterial | 12 months
  Frequency and gravity of unwanted Adverse Events linked to the procedure and\or the use of the biomaterial:
  O Inflammatory or allergic reaction to the tested product (VS and CRP before inclusion).
  * Non-union turned out and painful
  * Invalidating lumbar pain
  * Infection on the operated site
Evaluation of the pain | 12 months
  Evaluation of the pain with an analogical visual scale (EVA)
Quality of life evaluation | 12 years
  Quality of life evaluation by means of OSWESTRY and SF-36 scales

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles LE HUEC, PUPH, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- Unité d'Orthopédie-Traumatologie rachis II, Pellegrin, Bordeaux, France

REFERENCES:
- [Background] Anand N, Hamilton JF, Perri B, Miraliakbar H, Goldstein T. Cantilever TLIF with structural allograft and RhBMP2 for correction and maintenance of segmental sagittal lordosis: long-term clinical, radiographic, and functional outcome. Spine (Phila Pa 1976). 2006 Sep 15;31(20):E748-53. doi: 10.1097/01.brs.0000240211.23617.ae. PMID 16985443
- [Background] Battie MC, Videman T, Levalahti E, Gill K, Kaprio J. Genetic and environmental effects on disc degeneration by phenotype and spinal level: a multivariate twin study. Spine (Phila Pa 1976). 2008 Dec 1;33(25):2801-8. doi: 10.1097/BRS.0b013e31818043b7. PMID 19050586
- [Background] Battie MC, Videman T, Kaprio J, Gibbons LE, Gill K, Manninen H, Saarela J, Peltonen L. The Twin Spine Study: contributions to a changing view of disc degeneration. Spine J. 2009 Jan-Feb;9(1):47-59. doi: 10.1016/j.spinee.2008.11.011. PMID 19111259
- [Background] Carter JD, Swearingen AB, Chaput CD, Rahm MD. Clinical and radiographic assessment of transforaminal lumbar interbody fusion using HEALOS collagen-hydroxyapatite sponge with autologous bone marrow aspirate. Spine J. 2009 Jun;9(6):434-8. doi: 10.1016/j.spinee.2008.11.004. Epub 2008 Dec 25. PMID 19111510
- [Background] Chen Z, Zhao J, Liu A, Yuan J, Li Z. Surgical treatment of recurrent lumbar disc herniation by transforaminal lumbar interbody fusion. Int Orthop. 2009 Feb;33(1):197-201. doi: 10.1007/s00264-008-0531-1. Epub 2008 Mar 21. PMID 18357449
- [Background] el-Masry MA, Khayal H, Salah H. Unilateral transforaminal lumbar interbody fusion (TLIF) using a single cage for treatment of low grade lytic spondylolisthesis. Acta Orthop Belg. 2008 Oct;74(5):667-71. PMID 19058702
- [Background] Goyal N, Wimberley DW, Hyatt A, Zeiller S, Vaccaro AR, Hilibrand AS, Albert TJ. Radiographic and clinical outcomes after instrumented reduction and transforaminal lumbar interbody fusion of mid and high-grade isthmic spondylolisthesis. J Spinal Disord Tech. 2009 Jul;22(5):321-7. doi: 10.1097/BSD.0b013e318182cdab. PMID 19525786
- [Background] Houten JK, Post NH, Dryer JW, Errico TJ. Clinical and radiographically/neuroimaging documented outcome in transforaminal lumbar interbody fusion. Neurosurg Focus. 2006 Mar 15;20(3):E8. doi: 10.3171/foc.2006.20.3.9. PMID 16599424
- [Background] Jagannathan J, Sansur CA, Oskouian RJ Jr, Fu KM, Shaffrey CI. Radiographic restoration of lumbar alignment after transforaminal lumbar interbody fusion. Neurosurgery. 2009 May;64(5):955-63; discussion 963-4. doi: 10.1227/01.NEU.0000343544.77456.46. PMID 19404155
- [Background] Lauber S, Schulte TL, Liljenqvist U, Halm H, Hackenberg L. Clinical and radiologic 2-4-year results of transforaminal lumbar interbody fusion in degenerative and isthmic spondylolisthesis grades 1 and 2. Spine (Phila Pa 1976). 2006 Jul 1;31(15):1693-8. doi: 10.1097/01.brs.0000224530.08481.4e. PMID 16816765
- [Background] Rihn JA, Patel R, Makda J, Hong J, Anderson DG, Vaccaro AR, Hilibrand AS, Albert TJ. Complications associated with single-level transforaminal lumbar interbody fusion. Spine J. 2009 Aug;9(8):623-9. doi: 10.1016/j.spinee.2009.04.004. Epub 2009 May 30. PMID 19482519
- [Background] Rihn JA, Makda J, Hong J, Patel R, Hilibrand AS, Anderson DG, Vaccaro AR, Albert TJ. The use of RhBMP-2 in single-level transforaminal lumbar interbody fusion: a clinical and radiographic analysis. Eur Spine J. 2009 Nov;18(11):1629-36. doi: 10.1007/s00586-009-1046-1. Epub 2009 May 28. PMID 19475434
- [Background] Sasso RC, LeHuec JC, Shaffrey C; Spine Interbody Research Group. Iliac crest bone graft donor site pain after anterior lumbar interbody fusion: a prospective patient satisfaction outcome assessment. J Spinal Disord Tech. 2005 Feb;18 Suppl:S77-81. doi: 10.1097/01.bsd.0000112045.36255.83. PMID 15699810
- [Background] Schleicher P, Beth P, Ottenbacher A, Pflugmacher R, Scholz M, Schnake KJ, Haas NP, Kandziora F. Biomechanical evaluation of different asymmetrical posterior stabilization methods for minimally invasive transforaminal lumbar interbody fusion. J Neurosurg Spine. 2008 Oct;9(4):363-71. doi: 10.3171/SPI.2008.9.10.363. PMID 18939923
- [Background] Xiao Y, Li F, Chen Q. Transforaminal lumbar interbody fusion with one cage and excised local bone. Arch Orthop Trauma Surg. 2010 May;130(5):591-7. doi: 10.1007/s00402-009-0917-6. Epub 2009 Jun 30. PMID 19565252
- [Background] Xiao YX, Chen QX, Li FC. Unilateral transforaminal lumbar interbody fusion: a review of the technique, indications and graft materials. J Int Med Res. 2009 May-Jun;37(3):908-17. doi: 10.1177/147323000903700337. PMID 19589277
- [Background] Yan DL, Pei FX, Li J, Soo CL. Comparative study of PILF and TLIF treatment in adult degenerative spondylolisthesis. Eur Spine J. 2008 Oct;17(10):1311-6. doi: 10.1007/s00586-008-0739-1. Epub 2008 Aug 7. PMID 18685873